CLINICAL TRIAL: NCT00717262
Title: A Phase 1, Double-Blind, Placebo Controlled, Repeat-Dose Study of the Safety, Activity and Pharmacokinetics of HQK-1001 in Healthy Volunteers
Brief Title: Phase 1 Placebo Controlled Study of the Safety, Activity and Pharmacokinetics of HQK-1001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Susan Perrine, MD/ Chief Scientific Officer, HemaQuest Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HQP 2008-002
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
MeSH Terms: interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): HQK-1001
  Interventions: Drug: HQK-1001
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HQK-1001 — HQK-1001 (5, 10 or 15 mg/kg) capsules administered once a day, orally, for 14 days.
  Arms: 1
Drug: placebo — Matching placebo capsules administered once a day, orally, for 14 days.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety, activity and pharmacokinetics of a new investigational drug (HQK-1001) in healthy human volunteers. This study will also evaluate if there are differences in these parameters when HQK-1001 is administered in a fed versus a fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Between the ages of 18 and 45 years old
* Able and willing to give informed consent
* Able to comply with all study procedures
* If female, must not be of childbearing potential or must agree to use one or more of the following forms of contraception during screening and throughout the study: hormonal (i.e., oral, transdermal, implant or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD); vasectomized partner (6 months minimum); or abstinence
* Male subjects must also agree to use one or more of the above forms of birth control for either themselves or their partner, as appropriate, throughout the course of the study
* Not receiving medications within the 2 weeks before the first dose of study medication, except for multivitamins and contraception
* Complete blood count (CBC) with white blood cell (WBC) count hemoglobin, hematocrit, reticulocyte count and platelet count within normal range for the testing facility or not clinically significant
* Serum ferritin level > 50 ng/ml in Cohort 1
* Serum ferritin level > 30 mg/ml in Cohorts 2, 3, 4 and 5
* Serum chemistry values, coagulation tests and urinalysis values within the normal range for the testing facility or not clinically significant
* Negative urine test for substances of abuse including marijuana, cocaine, opiates, and methadone

Exclusion Criteria:

* Prior participation in HQP 2007-001
* Clinically significant abnormal vital signs
* Blood donation within 2 months of study medication administration
* Blood transfusion within 3 months of study medication administration
* An acute febrile illness or upper respiratory tract illness within 72 hours prior to administration of study medication
* Received another investigational agent within 4 weeks before administration of study medication
* Receiving any other investigational agent during this study
* Any acute or chronic disease (e.g., history of hepatitis B or C or HIV-1)
* Heart disease including an abnormal electrocardiogram, clinical significant, (ECG) or cardiac arrhythmia
* History of neurological disease, such as a seizure disorder
* Currently pregnant or breast feeding a child
* A smoker in the past 12 months
* Body Mass Index (BMI) >33 kg/m2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by (1) adverse events, (2) laboratory values (3) vital signs (4) physical exam | 41 days

SECONDARY OUTCOMES:
Pharmacokinetics assessed by plasma drug concentration levels | 15 days
Pharmacodynamics assessed by red blood cell production and induction of fetal hemoglobin | 41 days
Comparison of safety, PK and PD under fed versus fasting conditions | 41 days
Comparison of safety and PK when oral iron is administered with HQK-1001. | 41 days

CONTACTS AND LOCATIONS:
Overall Officials: Robin Downey, MD, Principal Investigator — Charles River Clinical Services Northwest
Locations (1):
- Charles River Clinical Services Northwest, Tacoma, Washington, United States